CLINICAL TRIAL: NCT03405272
Title: Recombinant Anti-EGFR Monoclonal Antibody（SCT200） in Patients With Chemotherapy- Refractory Wild Type RAS and BRAF Metastatic Colorectal Cancer
Brief Title: Safety and Efficacy of Recombinant Anti-EGFR Monoclonal Antibody in Patients With Wild-type RAS and BRAF mCRC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sinocelltech Ltd. (Industry)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCT200mCRCⅡ
Record Dates: First submitted 2018-01-11; First posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Full human anti-EGFR monoclonal antibody (SCT200); metastatic colorectal cancer （mCRC）
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Treated with recombinant anti-EGFR Monoclonal antibody（SCT200）until disease progression
Masking Description: Single Arm, Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- recombinant anti-EGFR monoclonal antibody（SCT200） (Experimental): Initially, 6.0mg/kg of SCT200 will be administered once a week for a maximum of 6 cycles. After 6 cycles, 8.0mg/kg of SCT200 will be administered every two weeks until disease progression.
  Interventions: Biological: Recombinant Anti-EGFR Monoclonal Antibody（SCT200）

INTERVENTIONS:
Biological: Recombinant Anti-EGFR Monoclonal Antibody（SCT200） — Experimental: recombinant anti-EGFR monoclonal antibody（SCT200） Recombinant Anti-EGFR Monoclonal Antibody（SCT200）. Initially, SCT200 6.0mg/kg will be administered at day 1 every week for a maximum of 6 cycles. After 6 cycles SCT200 8.0mg/kg will be administered at day 2 every weeks until disease progression.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of recombinant anti-EGFR Monoclonal antibody（SCT200）in patients with wild-type RAS and BRAF mCRC treated with fluorouracil, oxaliplatin and irinotecan after failure of standard therapy

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent and can understand and comply with the requirements of the study;
2. Men and women ≥ 18 years of age;
3. Life expectancy of longer than 3 months ( clinical assessment);
4. With an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1;
5. Have been diagnosed as mCRC verified histologically;
6. Patients treated with fluorouracil, oxaliplatin and irinotecan after failure of standard therapy. Disease progressed or developed non-tolerable toxicity after systemic chemotherapy：a. at least one treatment cycle should be completed, and maintenance therapy using one of the doublets is considered as the same line of therapy ; b. May have received adjuvant therapy for primary colorectal cancer provided that at least 6 months have elapsed from the time the adjuvant therapy was concluded and recurrent disease was documented;
7. RAS and BRAF wildtype status of primary colorectal cancer or related metastasis;
8. Adequate organ and marrow function as defined below:

   Absolute neutrophil count (ANC) greater than/equal to 1.5×l09/L; Platelets greater than/equal to 75×109/L; Hemoglobin greater than/equal to 80g/L; Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) less than/equal to 2.5 times IULN, or less than/equal to 5 times IULN if known liver metastases; Total bilirubin less than/equal to 1.5 within institutional upper limit of normal (IULN); Serum creatinine less than/equal to 1.5 times IULN; Electrolyte: magnesium greater than/equal to normal.
9. According to RECIST 1.1 , patients must have at least one measurable lesion that can be accurately assessed at baseline and is suitable for repeated assessment by CT, MRI. Longest diameter greater than/equal to10mm（CT scan slice thickness no greater than 5 mm）, a lymph node must be ≥15mm in short axis when assessed by CT scan.

Exclusion Criteria:

1. Patient with active brain metastasis or indicated for symptomatic treatment for brain metastasis, untreated with proper radiation therapy, showing clinical symptoms or symptom stable time less than 28 days;
2. Patients with other primary malignancies within the past 5 years except non-melanoma skin cancer, carcinoma in situ of cervix or prostatic intraepithelial neoplasia;
3. Patients who are allergic to analogue of SCT200 and/or its inactive ingredients;
4. Patients administrated EGFR target treatment including EGFR TKI agent or anti- EGFR monoclonal antibody;
5. Within 4 weeks, patients received anti-tumor drugs (such as chemotherapy, hormone therapy, immune therapy, the antibody therapy, radiotherapy) or research drugs, or patients with grade 2 or more adverse reaction caused by previous anti-tumor therapy(except alopecia or neurotoxicity grade 2 or less);
6. Patients are currently enrolled in other research devices or in research drugs, or less than 4 weeks from other research drugs or devices.
7. Patients received major surgery(such as need general anesthesia ) within 4 weeks , should recover from the injury associated with the surgery.
8. Patients treated with EPO, G-CSF or GM-CSF.
9. Patients who have clinically significant cardiovascular disease (defined as unstable angina pectoris, symptomatic congestive heart failure (NYHA, greater than II), uncontrollable severe arrhythmia);
10. Patients occurred myocardial infarction within 6 months.
11. Patients who have interstitial lung disease, such as interstitial pneumonia, pulmonary fibrosis, or CT or MRI reminder ILD .
12. Patients with clinical symptoms, required clinical intervention or stable time less than 4 weeks of serous cavity effusion (such as pleural effusion and ascites);
13. Patients with serious psychological or psychiatric disorders which may affect subject compliance in this clinical study;
14. Pregnant or lactating women, or women who planned to be pregnant within 6 months of treatment;
15. Patients who were not willing to accept effective contraceptive measures (including male or female subjects) during treatment and within 6 months after treatment;
16. Patients with active hepatitis B or active hepatitis C, etc. (for patients with a history of hepatitis B, whether treated or not, HBV DNA ≥104 or ≥ 2000IU/ml, HCV RNA≥15IU/ml); HIV antibody positive (if there is no clinical evidence suggesting that there may be HIV infection, there is no need to detect);
17. Patients with uncontrolled active infections before enrollment 2 weeks (except simple urinary tract infection or upper respiratory tract infection);
18. Patients have alcohol or drug addiction;
19. Inability to comply with study and/or follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2018-02-12 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 1 year
  The achievement of either a partial response (PR) or complete response (CR), according to RECIST 1.1 criteria

SECONDARY OUTCOMES:
Objective response rate - left side | 1 year
  The achievement of either a partial response (PR) or complete response (CR), left side mCRC patients treated by SCT200. according to RECIST 1.1 criteria
Best of response | 1 year
  Number of patients in each response category（CR, PR, SD, PD）, according to RECIST 1.1 criteria
Duration of response | 1 year
  Defined as the time from the date that the response criteria are first met to the date that progressive disease (PD) is objectively documented or death, whichever occurs first.
Disease control rate | 1 year
  The achievement of any a stableresponse（SD）, partial response (PR) or complete response (CR), according to RECIST 1.1 criteria
Time to response | 1 year
  Defined as the time from first dose of SCT200 to documentation of a response.according to RECIST 1.1 criteria
Progression free survival | 1 year
  Defined as time from first dose of SCT200 until first documentation of Progression or death, whichever comes first， according to RECIST 1.1 criteria
Overall survival | 1 year
  Defined as the time from first dose of SCT200 until death.

CONTACTS AND LOCATIONS:
Overall Officials: yuankai shi, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (21):
- China (21):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Cancer hospital Chinese academy of medical sciences, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The Sixth Affiliated Hospital Of Sun Yat-sen University, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital., Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Xiking Hospital, Xi'an, Shaanxi
  - Lin Yi Cancer Hospital, Linyi, Shandong
  - Zhongshan hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital Of Xinjiang Medical University, Ürümqi, Xinjiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang